CLINICAL TRIAL: NCT03535792
Title: The Efficacy Of Nalbuphine Versus Fentanyl As Additives To Bupivacaine In Spinal Anaesthesia For Internal FixationI Of Tibia
Brief Title: Nalbuphine Versus Fentanyl As Additives To Bupivacaine In Spinal Anaesthesia For Internal FixationI Of Tibia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Mohammad Hazem I. Ahmad Sabry, Lecturer of Anesthesia, University of Alexandria
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 050108393
Record Dates: First submitted 2018-05-12; First posted 2018-05-24 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Fentanyl; Nalbuphine

STUDY DESIGN:
Intervention Model Description: Group F:
  25 Patients will receive intrathecal injection of 2 ml of 0.5% hyperbaric bupivacaine plus 1 ml fentanyl (50μg).
  Group N:
  25 Patients will receive intrathecal injection of 2 ml of 0.5% hyperbaric bupivacaine plus 1ml nalbuphine hydrochloride (1.6 mg); (nalufin 20 mg in 1 ml ampoule, Amoun Pharmaceutical Co. Cairo, Egypt).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participant, care provider and outcome assessor will not be informed with the medication used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fentanyl/Hyperbaric Bupivacaine (Active Comparator): Group F:
  Patients will receive intrathecal injection of 2 ml of 0.5% hyperbaric bupivacaine plus 1 ml fentanyl (50μg) and will have Tibial internal fixation.
  Interventions: Drug: Fentanyl/Hyperbaric bupivacaine
- Nalbuphine/Hyerbaric Bupivacaine (Active Comparator): Group N:
  Patients will receive intrathecal injection of 2 ml of 0.5% hyperbaric bupivacaine plus 1ml nalbuphine hydrochloride (1.6 mg); (nalufin 20 mg in 1 ml ampoule, Amoun Pharmaceutical Co. Cairo, Egypt) and will have Tibial internal fixation.
  Interventions: Drug: Nalbuphine/Hyperbaric bupivacaine

INTERVENTIONS:
Drug: Fentanyl/Hyperbaric bupivacaine — Intrathecal Fentanyl/Hyperbaric bupivacaine and Tibial internal fixation.
  Other Names: Spinal Fentanyl/Hyperbaric bupivacaine
  Arms: Fentanyl/Hyperbaric Bupivacaine
Drug: Nalbuphine/Hyperbaric bupivacaine — Intrathecal Nalbuphine/Hyperbaric bupivacaine and Tibial internal fixation.
  Other Names: Spinal Nalbuphine/Hyperbaric bupivacaine
  Arms: Nalbuphine/Hyerbaric Bupivacaine

SUMMARY:
The Efficacy Of Nalbuphine Versus Fentanyl As Additives To Bupivacaine In Spinal Anaesthesia For Internal FixationI Of Tibia

DETAILED DESCRIPTION:
The Efficacy Of Nalbuphine Versus Fentanyl As Additives To Bupivacaine In Spinal Anaesthesia For Internal FixationI Of Tibia

INTRODUCTION Regional techniques, such as spinal anaesthesia may offer advantages over general anaesthesia including reduced stress response to surgery and analgesia extending into the postoperative period.(1,2) Adequate pain management to facilitate rehabilitation and to accelerate functional recovery after lower limb orthopedic surgery is essential to enable patients to resume normal activity as soon as possible.(3) To increase the duration of analgesia produced by local anesthetic, a number of adjuvants have been added through the central neuraxial route.(4) The profound segmental anti-nociception produced by neuraxial opioids in doses much smaller than would be required for comparable anti-nociception if administered systemically has made them very popular and effective in the treatment of many painful states.(5)The anti-nociception is also devoid of motor, sensory and autonomic blockade so there is no paralysis or hypotension. Furthermore, the availability of a specific opioid receptor antagonist naloxone to reverse their action when necessary has made the use of opioids more acceptable.(6) Opioids work in the intrathecal space by activating opioid- receptors in the dorsal gray matter of spinal cord, which modulates the function of afferent pain fibers.(7)Intrathecal and epidural narcotics seem to modulate pain primarily at the spinal cord rather than in the brain as do intravenous narcotics.(8) Site of action in the spinal cord may provide analgesia with less sedation, confusion and nausea, which are adverse effects associated with intravenous narcotics.(9) Various opioids have been used along with bupivacaine to prolong its effect, to improve the quality of analgesia and minimize the requirement of postoperative analgesics.(10,11) The main obstacles for optimal use of opioids are their side effects which include pruritis, nausea/ emesis, constipation, urinary retention, respiratory depression, undesirable sedation and the development of tolerance/ dependence. Though some side effects may be benign but others like respiratory depression can prove to be life threatening.(12-14) Nalbuphine is a semisynthetic opioid with mixed mu antagonist and kappa agonist properties. When used singly or in combination with other agents it has the potential to maintain or even enhance opioid based analgesia while simultaneously mitigating the common mu-opioid side effects. (15) Nalbuphine binds readily to both mu- and kappa-receptors. The binding of nalbuphine to mu receptors only serves to competitively displace other mu-agonists from the receptor, without itself displaying any agonist activity.(16)When nalbuphine binds to kappa-receptors, however, it has an agonist effect. Kappa-opioid receptors are distributed throughout brain and spinal cord involved in nociception. Nalbuphine binds avidly to kappa-receptors in these areas to produce analgesia. This pattern of binding and effects defines nalbuphine as a mixed agonist-antagonist.(17) Fentanyl, a lipophilic opioid has rapid onset of action, It does not tend to migrate intrathecally to the 4th ventricle in sufficient concentration to cause delayed respiratory depression.(18,19)

AIM OF THE WORK The aim of our study is to compare the effect of intrathecal nalbuphine versus intrathecal fentanyl as adjuvants to bupivacaine, as regard the intra-operative and post-operative analgesia, the hemodynamic stability, the onset of sensory/motor block and the duration of action in patients undergoing internal fixation of tibia.

PATIENTS This study will be carried out in El-Hadara University Hospital on sixty patients aged 18-50 years; belonging to American Society of Anesthesiologists (ASA) physical status I and II, scheduled for elective internal fixation of tibia, of expected duration less than 3 h, under subarachnoid block, this prospective study will be done in a double-blinded, randomized way.

Exclusion criteria:

* Patients with significant co-existing conditions such as hepatic, renal and cardiovascular diseases.
* Patients with contraindications to regional anesthesia like local infection or bleeding disorders.
* Patients with allergy to opioids, long-term opioids use, and a history of chronic pain.

After approval from the local ethical committee, a written consent will be obtained from each patient.

Patients will be randomly allocated into two groups according to intrathecal drug injected using closed envelope method.

Group F:

Patients will receive intrathecal injection of 2 ml of 0.5% hyperbaric bupivacaine plus 1 ml fentanyl (50μg).

Group N:

Patients will receive intrathecal injection of 2 ml of 0.5% hyperbaric bupivacaine plus 1ml nalbuphine hydrochloride (1.6 mg); (nalufin 20 mg in 1 ml ampoule, Amoun Pharmaceutical Co. Cairo, Egypt).

METHODS

1. Preoperative preparation:

   Preoperative screening of all patients including:
   * History taking.
   * Complete physical examination.
   * Laboratory investigation:

     * Complete blood picture (CBC)
     * Prothrombin time (PT), partial thromboplastin time (PTT), Prothrombin activity and INR.
     * Liver enzymes: Aspartate transaminase, Alanine transaminase.
     * Serum urea and creatinine.
     * Fasting blood sugar. Nothing per month in previous 6 hours.
2. Monitoring:

   All patients will be monitored by:
   * Electrocardiogram (ECG) for heart rate (beat/min).
   * Non-invasive arterial blood pressure: mean arterial blood pressure (MAP), systolic blood pressure (SAP) and diastolic arterial blood pressure (DAP).
   * Pulse oximeter for arterial oxygen saturation (SaO2).
3. Intraoperative procedure:

   * After securing intravenous (18G) access in the non-dominant hand, preloading with Ringer's solution 10 ml/kg in 15 min will be done.
   * Subarachnoid block will be performed with 3 ml of the study drug injected in L3/4 intervertebral space, using a 25 gauge Quincke spinal needle, in the sitting position, maintaining aseptic precautions, according to the standard institutional protocol.
   * The patients will be randomized using close envelope method equally into two groups according to the additive (fentanyl or nalbuphine), and all patients will receive the same amount of local anesthetic (2 ml 0.5% heavy bupivacaine).

   Thereafter, patients will be placed in the supine position for surgery, elevation of the head by a pillow and oxygen mask will be applied.

   Advanced equipment and drugs for resuscitation, airway management and ventilation will be ready.

   MEASUREMENTS 1. Hemodynamic parameters:
   * Patient heart rate and mean arterial blood pressure will be monitored and recorded at the following periods:
   * 5 minutes before the intrathecal injection.
   * At 2, 4, 6, 8 and 10 minutes after the injection.
   * Every 15 min until the patient will be moved to the post anaesthesia care unit (PACU).

     2. Assessment of sensory blockade:
   * The onset of sensory block is defined as the time in minutes to reach highest sensory level (20), it will be evaluated by ice at midclavicular level bilaterally every 2min for 15 min.
   * The duration of sensory block will be defined as the time it takes for sensory level to decrease to dermatomal level 12 measured from the highest sensory level evaluated by ice every 15 minutes. (21)
   * The maximal level of sensory block will be evaluated by 20 min after the completion of injection.

     3. Assessment of the motor block:
   * Onset time of motor block will be assessed immediately after sensory block assessment using modified Bromage scale.(22)

   Modified Bromage scale
   * The onset of motor block will be defined as the time from intrathecal injection to Bromage score 3 tested every 2min for 15 min. (23)
   * Duration of motor block will be evaluated every 15 minutes intraoperative from Bromage score 3 then every 30 minutes in the post anaesthesia care unit (PACU) until full recovery of motor function.
4. post operative analgesia:

   1. Duration of analgesia:

      * The duration of analgesia will be defined as the period from spinal injection to the first time when the patient complained of pain in the postoperative period.
      * Patients will be assessed using Visual analogue scale (VAS), in the immediate postoperative period, then every 2hours for the first 8hours, then every 6hours for the rest of the first 24hours.

      Visual analogue scale (VAS)

      - It ranges from 0 indicating no pain till 10 indicating severe intolerable pain with variable degrees of ascending pain in between.(24)
   2. Postoperative analgesic requirements:

      * The time of the first request analgesia will be recorded and treated by intramuscular diclofenac sodium (75mg) in a dose of 1mg/kg and repeated after 1 hour if needed up to 2 ampoules.
      * Paracetamol 1 g IV every 8 hours will be given for analgesia to all patients starting immediately postoperative (time zero).
      * Total dose of analgesic requirements will be calculated and elaborated statistically.
   3. Postoperative Complication:

Any complication will be recorded and managed such as hypotension, bradycardia, nausea, vomiting, pruritus, shivering and respiratory depression.

* Hypotension will be defined as systolic blood pressure less than 90mmHg and\or a decrease of more than 20% from baseline blood pressure. (25)
* Bradycardia will be defined as HR<50 beat\min.
* Respiratory depression will be defined as respiratory rate <10 breath\min.

ETHICS OF RESEARCH Prospective study: Informed consent will be taken from patients. In case of incompetent patients the informed consent will be taken from the guardians.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18-50 years
* American Society of Anesthesiologists (ASA) physical status I and II
* Scheduled for elective internal fixation of tibia, of expected duration less than 3 h, under subarachnoid block

Exclusion Criteria:

* Patients with significant co-existing conditions such as hepatic, renal and cardiovascular diseases.
* Patients with contraindications to regional anesthesia like local infection or bleeding disorders.
* Patients with allergy to opioids, long-term opioids use, and a history of chronic pain.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2017-11-04 (Actual); Primary Completion 2018-08-19 (Actual); Study Completion 2018-08-20 (Actual)

PRIMARY OUTCOMES:
Pain Postoperative | 24 hours
  VAS 0-10

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Hazem I Ahmad Sabry, MB,ChB MD, Principal Investigator — Alexandria University
Locations (1):
- Alexandria Faculty of Medicine, Alexandria, Egypt